CLINICAL TRIAL: NCT02511574
Title: Comparison Between Natural Progesterone and Vaginal Pessary for the Prevention of Spontaneous Preterm Birth in Pregnant Women With a Uterine Cervix Measuring 25 mm or Less in Length
Brief Title: Comparison Between Natural Progesterone and Vaginal Pessary for the Prevention of Spontaneous Preterm Birth
Acronym: PAP-C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Mario Henrique Burlacchini de Carvalho, Professor Doutor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 470.095
Record Dates: First submitted 2015-07-06; First posted 2015-07-30 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Preterm Labor; Premature Birth
Keywords: progesterone; uterine cervix; cervical pessary
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cervical pessary (Experimental): Patients with uterine cervical length ≤ 25 mm are randomized to use the cervical pessary or natural progesterone to compare their effectiveness in the reduction of preterm birth rates.
  Interventions: Device: cervical pessary
- natural progesterone (Active Comparator): Patients with uterine cervical length ≤ 25 mm are randomized to use the cervical pessary or natural progesterone to compare their effectiveness in the reduction of preterm birth rates.
  Interventions: Drug: natural progesterone

INTERVENTIONS:
Drug: natural progesterone
  Arms: natural progesterone
Device: cervical pessary
  Arms: cervical pessary

SUMMARY:
The aim of this study is to compare the effectiveness between the cervical pessary and the natural progesterone in reduction of preterm birth rates in pregnant women with a uterine cervical length of 25 mm or less evaluated by transvaginal ultrasonography.

DETAILED DESCRIPTION:
Preterm birth is the leading cause of perinatal morbidity and mortality. The rates of spontaneous premature labor have not changed much during the past 10 years. A significant decrease in mortality and morbidity of premature babies will only be possible if women at risk of spontaneous preterm birth are accurately identified and administered preventive therapies. Ultrasonographic measurement of the cervix between 20 and 24 weeks of gestation can improve the identification of both women with single pregnancies and those with twin pregnancies at risk. Asymptomatic women with a short uterine cervix (25 mm or less) are at increased risk of spontaneous premature labor.

The prophylactic use of progesterone during the early phase of pregnancy in women with a history of preterm birth and those with a short cervix can prevent preterm birth.

The cervical pessary is a device used also for the prevention of preterm birth. Vaginal infections are also important causes of preterm birth. There are not many studies about the vaginal microbiome in pregnant women.

Measurement of cervical length is used as a screening test because it is inexpensive, has a short learning curve, and is well tolerated by patients. In addition, placement and removal of the pessary is an easy, accessible, and noninvasive procedure. The results on the concentration of omega 3 and preterm birth are still conflicting.

The aim of this study is to compare the effectiveness of the cervical pessary and the natural progesterone in reduction of preterm birth rates in pregnant women with a uterine cervix measuring 25 mm or less in length as evaluated by transvaginal ultrasonography, assess whether there is a relationship between maternal plasma concentration of omega 3 and preterm birth, and compare the microbiome in these women.

Methods: A prospective randomized controlled trial including pregnant women at the time of morphological ultrasound between 20 and 23 weeks and 6 days of pregnancy. Pregnant women in this gestational age with cervical length of 25 mm or less will be randomized between the conduct and the inclusion of progesterone vaginal pessary. In patients of both groups vaginal discharge sample will be collected at the time of randomization.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 20 weeks and 23 weeks and 6 days
* singleton pregnancies

Exclusion Criteria:

* fetal death at randomization
* major structural or chromosomal abnormality
* cervical cerclage in the current pregnancy
* preterm rupture of membranes diagnosed before randomization

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Spontaneous preterm birth before 34 weeks of gestational age | before 34 weeks of gestation
  All births that occurred before 34 weeks of gestation were included, excluding iatrogenic births (medically indicated).

SECONDARY OUTCOMES:
Overall preterm birth before 37, 34, 32 and 30 weeks of gestational age | before 37, 34, 32 and 30 weeks of gestation
  All births (spontaneous and iatrogenic) that occurred before 37, 34, 32 and 30 weeks of gestation were included.
Spontaneous preterm birth before 37, 32 and 30 weeks of gestational age | before 37, 32 and 30 weeks of gestation
  All births that occurred before 37, 32 and 30 weeks of gestation were
Adverse neonatal events | Neonatal period (up to 27 days after birth)
  Intraventricular hemorrhage, respiratory distress syndrome, retinopathy of prematurity and necrotizing enterocolitis
The need of neonatal special care | Neonatal period (up to 27 days after birth)
  admission to neonatal intensive care unit [NICU], mechanical ventilation, phototherapy, treatment for sepsis and blood transfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, Brazil